CLINICAL TRIAL: NCT01275313
Title: RCT on Wheeled Mobility for Preventing Pressure Ulcers
Brief Title: Wheeled Mobility for Preventing Pressure Ulcers
Acronym: RCT-WC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Brienza, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO09120362; R01HD041490 (NIH)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Mobility Limitation
Keywords: Pressure ulcers; wheelchairs; wheelchair functional capacity; custom-fitted wheelchair
MeSH Terms: conditions — Mobility Limitation; Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custom-Fitted Lightweight Wheelchair & Cushion (Experimental): Receive a new custom-fitted lightweight wheelchair, skin protection cushion and wheelchair skills training
  Interventions: Device: Lightweight wheelchair
- Cushion Only (Other): Receive a skin protection cushion and wheelchair training, but remain in facility-issued wheelchair
  Interventions: Device: Skin Protection Cushion

INTERVENTIONS:
Device: Lightweight wheelchair — Seating and wheeled mobility assessment and fitting of a lightweight wheelchair
  Arms: Custom-Fitted Lightweight Wheelchair & Cushion
Device: Skin Protection Cushion — Seating assessment and provision of a cushion meeting CMS code for Skin Protection wheelchair cushion
  Arms: Cushion Only

SUMMARY:
The proposed clinical trial is aimed at demonstrating the important role wheelchairs play in preventing pressure ulcers (bed sores). Although most pressure ulcers can be prevented, they are common in nursing home settings because their causes are difficult to identify. This clinical trial will guide practitioners toward improving preventive care practices by demonstrating how to effectively apply wheelchair and seat cushion technology.

DETAILED DESCRIPTION:
Pressure ulcers are a significant healthcare problem for the growing number of nursing home residents in the United States and around the world. Pressure ulcers diminish quality of life, exact a devastating loss of function, increase the risk of death in geriatric populations and raise healthcare costs. Costs for the management of pressure ulcers in the US likely exceeds $6.4 billion annually, with a prevalence of approximately 12% in the high risk LTC population. A previous clinical trial at the University of Pittsburgh studied the effects of seat cushions on pressure ulcer incidence and found that when a skin protection seat cushion is used with a properly fitted wheelchair there is a significant reduction in incidence. The data led the investigators to question whether having a properly fitted wheelchair also has a significant effect on pressure ulcer incidence. This clinical trial investigate this question by randomizing subjects into a control group that receives a skin protection cushion and wheelchair training for use in their facility supplied wheelchair, or a treatment group that receives a skin protection cushion, wheelchair training and a new custom-fitted wheelchair. We expect that the treatment group will have a lower incidence of pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female nursing home resident 60 years of age and older
2. A Braden score of less than or equal to 18
3. A combined Braden Activity and Mobility Subscale score less than or equal to 5
4. Absence of ischial and sacral area pressure ulcers (see definition of pressure ulcer)
5. A tolerance for total daily wheelchair sitting time of greater than or equal to 6 hours (not continuous)
6. Ability to accommodate seating and positioning needs with the wheelchair selected for use in this study (Breezy Ultra 4)
7. Informed written consent

Exclusion Criteria:

1. Body weight exceeding 250 lbs.
2. Hip width exceeding 20 in.
3. Wheelchair seating requirements for additional head support, seat depth > 20 inches, elevated leg rests or severe orthopedic deformities of the pelvis, lower extremities or back that exceed the accommodating capability of the Breezy Ultra 4 wheelchair.
4. Current use of any cushioning material(s) other than a standard cushion, a folded pad, or a pillow (standard cushion as defined by HCPCS code for Standard Cushions, i.e., non-skin protection cushion)
5. Current use of a HCPCS code K0004 wheelchair

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Brienza, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Brienza D, Kelsey S, Karg P, Allegretti A, Olson M, Schmeler M, Zanca J, Geyer MJ, Kusturiss M, Holm M. A randomized clinical trial on preventing pressure ulcers with wheelchair seat cushions. J Am Geriatr Soc. 2010 Dec;58(12):2308-14. doi: 10.1111/j.1532-5415.2010.03168.x. Epub 2010 Nov 10. PMID 21070197
- [Derived] Brienza DM, Karg PE, Bertolet M, Schmeler M, Poojary-Mazzotta P, Vlachos H, Wilkinson D. A Randomized Clinical Trial of Wheeled Mobility for Pressure Injury Prevention and Better Function. J Am Geriatr Soc. 2018 Sep;66(9):1752-1759. doi: 10.1111/jgs.15495. Epub 2018 Aug 10. PMID 30094810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Custom-Fitted Lightweight Wheelchair & Cushion | Cushion Only
Started | 127 | 131
Completed | 102 | 79
Not Completed | 25 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom-Fitted Lightweight Wheelchair & Cushion | Cushion Only | Total
Number analyzed (Participants) | 127 | 131 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 89.0 (8.7) | 89.1 (9.2) | 89.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 105 | 202
  Male | 30 | 26 | 56
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (5.2) | 26.9 (5.8) | 26.5 (5.5)
Incontinent [Count of Participants; unit: Participants] | 102 | 95 | 197
Previous history of pressure injury [Count of Participants; unit: Participants] | 27 | 17 | 44
Patient alert and oriented [Count of Participants; unit: Participants] | 114 | 116 | 230
Ambulation Distance [Count of Participants; unit: Participants]
  0 ft | 63 | 77 | 140
  <= 10 ft | 28 | 22 | 50
  >10 ft | 36 | 31 | 67
  Unknown | 0 | 1 | 1
Sensation [Count of Participants; unit: Participants]
  Normal | 96 | 88 | 184
  Diminished/Questionable | 26 | 31 | 57
  Absent | 1 | 0 | 1
  Unknown | 4 | 12 | 16
Scoliosis [Count of Participants; unit: Participants]
  Neutral | 89 | 83 | 172
  Flex deformity | 23 | 23 | 46
  Fixed deformity | 11 | 13 | 24
  Unknown | 4 | 12 | 16
Kyphosis [Count of Participants; unit: Participants]
  Neutral | 26 | 26 | 52
  Flex deformity | 65 | 64 | 129
  Fixed deformity | 32 | 29 | 61
  Unknown | 4 | 12 | 16
Lordosis [Count of Participants; unit: Participants]
  Neutral | 123 | 119 | 242
  Unknown | 4 | 12 | 16
Pelvic tilt [Count of Participants; unit: Participants]
  Neutral | 32 | 35 | 67
  Flex deformity | 64 | 62 | 126
  Fixed deformity | 27 | 22 | 49
  Unknown | 4 | 12 | 16
Pelvic Rotation [Count of Participants; unit: Participants]
  Neutral | 97 | 87 | 184
  Flex deformity | 24 | 28 | 52
  Fixed deformity | 2 | 4 | 6
  Unknown | 4 | 12 | 16
Pelvic Obliquity [Count of Participants; unit: Participants]
  Neutral | 102 | 93 | 195
  Flex deformity | 18 | 21 | 39
  fixed deformity | 3 | 5 | 8
  Unknown | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Incidence of a Sitting-induced Pressure Ulcer
Description: Skin assessments for incidence of sitting-induced pressure ulcers will occur once per week until the occurrence of a pressure ulcer or 182 days
Time Frame: 182 days
Measure: Count of Participants; unit: Participants
Arm/Group | Custom-Fitted Lightweight Wheelchair & Cushion | Cushion Only
Number analyzed (Participants) | 102 | 89
Participants
  Seating surface pressure injury | 19 | 15
  26 weeks since initiation of seating intervention | 75 | 69
  Death | 8 | 5
Statistical Analysis 1: Comparison: Custom-Fitted Lightweight Wheelchair & Cushion vs Cushion Only; Null hypothesis: At-risk nursing home residents provided with an individually-configured manual lightweight wheelchair and skin protection cushion have the same incidence of pressure injury development compared to individuals using a facility-provided manual wheelchair modified with a skin protection cushion and related adjustments; Test type: Equivalence — Power calculation: To determine a difference of 20% in the control group and 10% in the treatment group with 80% power, 440 participants would be needed; p = 0.77, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Custom-Fitted Lightweight Wheelchair & Cushion | Cushion Only
All-Cause Mortality (participants affected / at risk) | 8/127 | 5/131
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/131
Other Adverse Events (participants affected / at risk) | 0/127 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No